CLINICAL TRIAL: NCT01663233
Title: A Randomized, 8-week, Double-blind, Parallel-group, Active-controlled, Multicenter Study to Evaluate the Efficacy and Safety of the Combination of LCZ696 200 mg + Amlodipine 5 mg in Comparison With Amlodipine 5 mg in Patients With Essential Hypertension Not Adequately Responsive to Amlodipine 5 mg Monotherapy Treatment
Brief Title: Efficacy and Safety of LCZ696 200 mg + Amlodipine 5 mg in Comparison With Amlodipine 5 mg in Hypertensive Patients Not Responding to Amlodipine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLCZ696A2319
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; High blood pressure
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCZ696 and amlodipine (Experimental): Participants, first treated with 5 mg of amlodipine for 4 weeks to determine if they were not adequately responding to amlodipine (had an office msSBP ≥145 mmHg and <180 mmHg) and who met all inclusion and exclusion criteria), were randomized to receive 200mg of LCZ696 in combination with 5 mg of amlodipine for 8 weeks.
  Interventions: Drug: LCZ696; Drug: Amlodipine
- Amlodipine (Active Comparator): Participants, first treated with 5 mg of amlodipine for 4 weeks to determine if they were not adequately responding to amlodipine (had an office msSBP ≥145 mmHg and <180 mmHg) and who met all inclusion and exclusion criteria), were randomized to receive 5 mg of amlodipine and placebo to LCZ696 for 8 weeks.
  Interventions: Drug: Amlodipine; Drug: Placebo

INTERVENTIONS:
Drug: LCZ696 — LCZ696 will use tablets available at a strength of 200mg. Patients will be instructed to take the prescribed medication once a day.
  Arms: LCZ696 and amlodipine
Drug: Amlodipine — Amlodipine will use tablets available at a strength of 5 mg. Patients will be instructed to take the prescribed medication once a day.
Drug: Placebo — Matching placebo to LCZ696
  Arms: Amlodipine

SUMMARY:
This study will assess whether LCZ696 when used in combination with amlodipine will provide greater BP lowering benefit compared to amlodipine alone in Asian hypertensive patients not adequately responsive to amlodipine therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients must give written informed consent and have a diagnosis of hypertension:

Untreated patients must have an msSBP ≥ 150 mmHg and < 180 mmHg at both Visit 1 and Visit 101. Pre-treated patients must have an msSBP ≥ 145 mmHg and < 180 mmHg after wash out at Visit 101. All patients must have an office msSBP ≥ 145 mmHg and < 180 mmHg at the completion of the 4-week run-in epoch (at the randomization visit (Visit 201).

Patients must successfully complete ABPM and pass technical requirements at Visit 201.

Exclusion Criteria:

Malignant or severe hypertension (grade 3 of WHO classification; msDBP ≥110 mmHg and/or msSBP ≥ 180 mmHg).

History of angioedema, drug-related or otherwise. History or evidence of a secondary form of hypertension. Transient ischemic cerebral attack (TIA) during the 12 months prior to Visit 1 or any history of stroke.

History of myocardial infarction, coronary bypass surgery or PCI during the 12 months prior to Visit 1

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- China (4):
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Japan (7):
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Kunitachi, Tokyo
  - Novartis Investigative Site, Shibuya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Malaysia (2):
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Philippines (4):
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Quezon City
  - Novartis Investigative Site, Valenzuela
- South Korea (5):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Koyang, Kyunggi
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Daegu
- Taiwan (3):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC

RESULTS

PARTICIPANT FLOW:
Groups:
- LCZ696 and Amlodipine: Participants, first treated with 5 mg of amlodipine for 4 weeks to determine if they were not adequately responding to amlodipine (an office msSBP ≥145 mmHg and <180 mmHg) and who met all inclusion and exclusion criteria), were randomized to receive 200mg of LCZ696 in combination with 5 mg of amlodipine for 8 weeks.
- Amlodipine: Participants, first treated with 5 mg of amlodipine for 4 weeks to determine if they were not adequately responding to amlodipine (an office msSBP ≥145 mmHg and <180 mmHg) and who met all inclusion and exclusion criteria), were randomized to receive 5 mg of amlodipine and placebo to LCZ696 for 8 weeks.
Period: Overall Study
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Started | 130 | 136
Completed | 126 | 129
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Deviation | 1 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 and Amlodipine | Amlodipine | Total
Number analyzed (Participants) | 130 | 136 | 266
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.4 (9.31) | 55.5 (9.43) | 55.4 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 61 | 110
  Male | 81 | 75 | 156

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Systolic Blood Pressure (maSBP)
Description: The change in mean 24 hour ambulatory systolic blood pressure (maSBP) from baseline to end of the study (week 8) in the 2 groups was measured. A greater reduction from baseline in the LCZ696 group indicates a positive treatment effect.
Time Frame: 8 weeks
Population: FAS: This set included all randomized participants who received at least one dose of study medication. Among the 266 Full Analysis Set (FAS) participants, 251 participants (123 participants in the LCZ696 + amlodipine group and 128 participants in the amlodipine group) had eligible ABPM at both baseline and endpoint.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Number analyzed (Participants) | 123 | 128
mmHg | -13.93 (0.56) | -0.82 (0.56)

2. Secondary Outcome: Change in Mean 24-hour ABPM Diastolic Blood Pressure (maDBP)
Description: The change in mean 24 hour maDBP from baseline to end of the study was measured. A reduction from baseline indicates a positive treatment effect.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Number analyzed (Participants) | 123 | 128
mmHg | -8.03 (0.38) | -0.33 (0.37)

3. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: The change in the patient's msSBP from baseline to end of the study was measured. A reduction from baseline indicates a positive treatment effect.
Time Frame: 8 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Number analyzed (Participants) | 130 | 136
mmHg | -19.60 (1.35) | -9.34 (1.33)

4. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: The change in the patient's msDBP from baseline to end of the study was measured. A reduction from baseline indicates a positive treatment effect.
Time Frame: 8 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Number analyzed (Participants) | 130 | 136
mmHg | -9.22 (0.83) | -3.96 (0.82)

5. Secondary Outcome: Change in Sitting Pulse Pressure (PP)
Description: The change in the patient's mean sitting PP from baseline to end of the study was measured. Pulse pressure measures the difference in mean sitting systolic blood pressure and mean sitting diastolic blood pressure.
Time Frame: 8 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Number analyzed (Participants) | 130 | 136
mmHg | -10.31 (0.90) | -5.46 (0.89)

6. Secondary Outcome: Number of Participants Achieving Systolic and Diastolic Blood Pressure Control (< 140/90 mmHg)
Description: The number of participants achieving a systolic and diastolic blood pressure < 140/90 mmHg was measured. This outcome measure shows how well a given blood pressure treatment can achieve a given blood pressure target or goal. Participants who achieved the target blood pressure were determined based on the mean SBP and DBP measurements taken at the end of the study. If the participants' BP measurement was below the above target, they were considered to have successful blood pressure control.
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Number analyzed (Participants) | 130 | 136
Participants | 89 | 46

7. Secondary Outcome: Number of Participants Achieving Successful Response in msSBP (< 140 mmHg or a Reduction ≥ 20 mmHg From Baseline)
Description: The number of participants who achieved successful treatment response in the msSBP of < 140mmHg or a reduction ≥ 20 mmHg from baseline after completing study treatment was measured. Participants who achieved either of the above targets were deemed as a having a successful response.
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Number analyzed (Participants) | 130 | 136
Participants | 98 | 53

8. Secondary Outcome: Number of Participants Achieving Successful Response in msDBP (< 90 mmHg or a Reduction ≥ 10 mmHg From Baseline)
Description: The number of participants who achieved successful treatment response in msDBP of < 90mmHg or a reduction ≥ 10mmHg from baseline after completing study treatment was measured. Participants who achieved either of the above targets were deemed as having a successful response.
Time Frame: 8 weeks of treatment
Population: FAS
Measure: Number; unit: Participants
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Number analyzed (Participants) | 130 | 136
Participants | 112 | 95

9. Secondary Outcome: Number of Participants With Adverse Event
Description: Participants were monitored for adverse events, serious adverse events and death.
Time Frame: 8 weeks
Population: Safety Set: The safety set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Number analyzed (Participants) | 130 | 136
Participants
  Adverse Events (serious and non-serious) | 26 | 29
  Serious Adverse Events | 0 | 0
  Deaths | 0 | 0

ADVERSE EVENTS:
Arm/Group | LCZ696 and Amlodipine | Amlodipine
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/136
Other Adverse Events (participants affected / at risk) | 13/130 | 19/136
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 and Amlodipine (N=130) | Amlodipine (N=136)
NASOPHARYNGITIS (Infections and infestations) | 5 | 5
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 5
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 5
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 4
DIZZINESS (Nervous system disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.